CLINICAL TRIAL: NCT01953094
Title: The Overlooked Population at Risk for AIN: Women With High-grade Lower Genital Tract Dysplasia or Cervical Cancer.
Brief Title: Overlooked Population at Risk for AIN.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Danielle Vicus, Surgical Oncologist in Gynecology Site Group, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GYNEOCC 1
Record Dates: First submitted 2013-08-26; First posted 2013-09-30 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: High Grade Cervical Dysplasia; Cervical Cancer
Keywords: Cervical
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anal Screening Pap Smear - Negative (Other): Anal Pap Smear with no High Resolution Anoscopy
  Interventions: Procedure: Screening Anal Pap Smear - No High Resolution Anoscopy
- Anal Pap Smear - Positive Result - High Resolution Anoscopy (Other): Patient who have a positive anal pap smear will go on to have a high resolution anoscopy.
  Interventions: Procedure: Screening Anal Pap Smear - With High Resolution Anoscopy

INTERVENTIONS:
Procedure: Screening Anal Pap Smear - No High Resolution Anoscopy
  Arms: Anal Screening Pap Smear - Negative
Procedure: Screening Anal Pap Smear - With High Resolution Anoscopy
  Arms: Anal Pap Smear - Positive Result - High Resolution Anoscopy

SUMMARY:
The purpose of this study is to determine the possibility and compliance of performing anal Pap smear and Human Papilloma Virus (HPV) DNA testing on women with high grade lower genital tract dysplasia or cervical cancer and determining the prevalence of anal dysplasia in this population using a high-resolution anoscopy (HRA). In addition, it is being done to potentially develop screening, diagnostic and treatment protocol for anal dysplasia in women with high-grade lower genital tract dysplasia or cervical cancer.

DETAILED DESCRIPTION:
Anal cancer incidence is increasing and although women compose more than half of all cases and those with HPV related lower genital tract dysplasia/malignancy have an even greater risk screening is currently not recommended. We therefore propose performing a prospective cohort study to determine the prevalence of anal dysplasia in women with high-grade lower genital tract dysplasia using high-resolution anoscopy HRA. This will then potentially lead to the development of a screening, diagnosis and treatment schema that can be implemented in all women with high-grade lower genital tract dysplasia. This study can potentially have a high impact on health delivery in women at high risk for anal cancer as this can transform the current treatment of anal cancer to a preventive screening program. This can later be implemented throughout Ontario and in all centers that treat women with cervical dysplasia.

The incidence of anal intraepithelial neoplasm (AIN also known as anal cancer) has increased in Ontario over the last 20 years. Two-thirds of the cases are found in women. The average time between diagnosis of anal cancer and previous cervical dysplasia or cancer is approximately 20 years. This study is giving the opportunity to detect and treat pre-invasive lesions and potentially prevent the development of anal cancer. Currently, no screening, diagnosis or treatment recommendation for anal dysplasia found in women with high-grade lower genital tract dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 40 years old
* Previous or current high grade cervical dysplasia or cervical cancer

Exclusion Criteria:

* Women ≥ 40 years old because the median time between the diagnosis of anal cancer and previous cervical cancer is approximately 20 years.
* chemotherapy or radiation therapy within the last 6 months

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2014-10; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Prevalence | Screening and up to 24 weeks.
  Prevalence of anal dysplasia in women with high grade cervical dysplasia or cervical cancer. Calculated at screening all women with cervical dysplasia or cancer and performing high-resolution anoscopy on those diagnosed with dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Daniell Vicus, MD, Principal Investigator — Odette Cancer Centre
Locations (1):
- Odette Cancer Centre, Toronto, Ontario, Canada